CLINICAL TRIAL: NCT06454708
Title: An Open Phase I Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Single Dose and Repeat Dose Topical Administrations of Clascoterone Cream, 1% in Healthy Chinese Adult Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability of Clascoterone Cream 1% in Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Sunshine Mandi Pharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LWY23090P
Record Dates: First submitted 2024-05-31; First posted 2024-06-12 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clascoterone Cream 1% (Experimental)
  Interventions: Drug: Clascoterone Cream 1%

INTERVENTIONS:
Drug: Clascoterone Cream 1% — Clascoterone Cream 1% (Winlevi) is indicated for the topical treatment of acne vulgaris in patients 12 years of age and older.

SUMMARY:
The primary objective of this study is to determine the pharmacokinetics (PK) of Clascoterone Cream, 1% after single dose and repeat dose topical administrations in healthy Chinese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adult subjects, male or female;
* 18-45 years of age (18 years old and 45 years old are inclusive, on the day of signing the written informed consent);
* Males should be ≥50.0 kg females should be ≥45.0 kg, respectively, and their body mass index [BMI = weight (kg)/height2 (m2)] should be within the range of 19.0 to 28.0 kg/m2 (including critical value);
* Female subjects of childbearing potential or male subjects whose partners are of childbearing potential should agree and be able to use effective contraception from the time of signing the written informed consent to within 3 months after the last dosing (see Appendix 2 for details);
* Subjects should be able to communicate well with the investigator and complete the study as per the protocol; subjects should be fully informed about the study and sign a written informed consent voluntarily.

Exclusion Criteria:

* Subject has a previous history of chronic or serious disease;
* Subject who has undergone major surgical procedure or procedure affecting drug absorption, distribution, metabolism, or excretion within 6 months prior to screening, or plans to undergo surgery during the study;
* Subject has a history of drug abuse and drug dependence;
* Subject who has received any medication prior to screening;
* Subject has previous allergies or has allergic symptoms;
* Subject has skin damages;
* Subject who has consumed alcohol regularly;
* Subject has positive testing result of drug abuse and narcotics screening ;
* Subject who has consumed excessive of strong tea, coffee, or caffeine-containing beverages;
* Subject who has been addicted to smoking;
* Subject who has intake of grapefruit-rich beverages or foods;
* Subject who has participated in a clinical study with another drug or device and has used the drug or device prior to screening
* Subject who has donated blood or bled heavily , or received a blood transfusion or used blood products; or who plans to donate blood or blood components;
* Subject has abnormal physical examination result at screening, or abnormal result of vital signs, or abnormal ECG findings;
* Subject has abnormal and clinically significant results of clinical laboratory tests;
* Subject who is a pregnant or lactation woman or has positive pregnancy test result;
* Subject who is unable to follow a uniform diet;
* Subject who has difficulty in collecting blood, has a history of needle and blood fainting or cannot tolerate venipuncture;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Time to maximum plasma concentration (Tmax) | Day 1
  Time to maximum plasma concentration
Maximum plasma concentration (Cmax) | Day 1
  Maximum plasma concentration
Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration (AUC0-t) | Day 1
  Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration
Time to maximum plasma concentration (Tmax) | Day 7
  Time to maximum plasma concentration
Maximum plasma concentration at steady state (Cmax,ss) | Day 7
  Maximum plasma concentration at steady state
Minimum plasma concentration at steady state (Cmin,ss) | Day 7
  Minimum plasma concentration at steady state

SECONDARY OUTCOMES:
AEs and SAEs | Day 7
  Incidence and severity of all adverse events (AEs) and serious adverse events (SAEs), and their relevance with the investigational drug.
Temperature | Day 7
  Incidence of abnormal clinically significant temperature results.
Pulse rate | Day 7
  Incidence of abnormal clinically significant pulse rate results.
Blood pressure | Day 7
  Incidence of abnormal clinically significant blood pressure results.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, London, China

IPD SHARING:
Plan to Share IPD: No